CLINICAL TRIAL: NCT03351933
Title: A Prospective, Open-Label, Single-Arm Clinical Trial to Assess the Anti-Hepatitis A Virus (HAV) Antibody Levels, Pharmacokinetics, and Safety of a Single Intramuscular Dose of a Polyvalent Human Immune Globulin in HAV Seronegative Healthy Subjects
Brief Title: Anti-Hepatitis A Virus, Pharmacokinetics, and Safety of Immune Globulin (Human)
Acronym: GamaSTAN
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Grifols Therapeutics LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: GC1703
Record Dates: First submitted 2017-11-20; First posted 2017-11-24 (Actual); Results first posted 2019-07-30 (Actual); Last update posted 2019-07-30 (Actual); Status verified 2019-07

CONDITIONS: Anti-Hepatitis A Antibody Levels in Heathy Subjects
MeSH Terms: interventions — gamma-Globulins; Immunoglobulins, Intravenous

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Immune Globulin (Human) GamaSTAN (Experimental): The healthy subjects received a single IM dose of GamaSTAN (0.2 mL/kg), followed by a PK sampling period of 150 days.
  Interventions: Biological: Immune Globulin (Human)

INTERVENTIONS:
Biological: Immune Globulin (Human) — A single 0.2 mL/kg IM injection of Immune Globulin (Human) (GamaSTAN) was administered in healthy subjects.
  Other Names: GamaSTAN

SUMMARY:
This was a single center, open-label, single-arm study in which approximately 28 Hepatitis A virus (HAV)-seronegative healthy subjects were enrolled. There was a screening period of up to 28 days during which subjects were screened for enrollment in the study.

Healthy subjects received a single intramuscular (IM) dose of GamaSTAN (0.2 mL/kg), followed by a pharmacokinetic (PK) sampling period of 150 days (approximately 5 half-lives). The protective levels of anti-HAV antibodies were assessed up to 60 days after the administration of GamaSTAN. A PK curve was obtained during the PK sampling period.

DETAILED DESCRIPTION:
This was a single center, open-label, single-arm study design, in which approximately 28 subjects received the same study treatment (0.2 mL/kg dose via IM injection). There was no reference therapy in this study.

The study was explained to each subject prior to the subject providing written informed consent. All subjects were screened to ensure that all the inclusion criteria and none of the exclusion criteria were met.

A sufficient number of healthy male and female subjects were qualified by screening assessments and procedures for reporting to the clinical site on Day -1. The healthy subjects received a single IM dose of GamaSTAN (0.2 mL/kg) on Day 1. Subjects were discharged from the clinic on Day 2, following the scheduled assessments and procedures, and returned to the clinical site for the remaining ambulatory PK samples and safety monitoring, and again for the final visit (Day 150).

The total duration of study participation for subjects who completed the study were approximately 178 days.

ELIGIBILITY:
Inclusion Criteria:

1. Male subjects from 18 to 55 years of age, inclusive, or female subjects from 18 to 65 years of age, inclusive
2. Subjects with a body mass index (BMI) of 18.5 to 29.9 kg/m2
3. Body weight greater than or equal to 50 kg at screening
4. Subjects willing and able to provide written informed consent
5. Subjects in good health in the judgment of the Investigator, as determined by medical history, physical examination, vital signs, ECG and laboratory assessments
6. A female study subject must meet one of the following criteria:

   1. If a female of childbearing potential - agrees to use one of the accepted contraceptive regimens from at least 30 days prior to study treatment administration and during the entire study duration. An acceptable method of contraception includes one of the following:

      * Abstinence from heterosexual intercourse (i.e. when abstinence is the preferred and usual lifestyle of the subject; periodic abstinence is not acceptable)
      * Non-estrogen containing hormonal contraceptives (birth control pills, injectable/implant/insertable hormonal birth control products, transdermal patch)
      * Intrauterine device without hormones
      * Condom with spermicide
      * Diaphragm or cervical cap with spermicide
      * Vasectomized partner (minimum 6 months since vasectomy prior to study treatment administration)
   2. If a female of non-childbearing potential - should be surgically sterile (i.e. has undergone complete hysterectomy, bilateral oophorectomy, or tubal ligation) or in a menopausal state (at least 1 year without menses prior to study treatment administration)
7. A male study subject must agree to use one of the accepted contraceptive regimens during the entire study duration;

   * Abstinence from heterosexual intercourse
   * Female partner with condom with spermicide used by male study subject
   * Female partner of non-childbearing potential
   * Male sterilization (if proof of sterilization is not provided, the subject must agree to use one of the above accepted contraceptive methods)
8. A male study subject must agree not to impregnate a female or donate sperm during the entire study duration

Exclusion Criteria:

1. Subject vaccinated against HAV, as documented the in medical history at the screening visit
2. Subject with positive anti-HAV antibodies in blood sample at the screening visit
3. Subject who previously received any type of IG, including HAV IG within the past 12 months prior to study treatment administration
4. Subject with prolonged International Normalized Ratio (INR) or activated partial thromboplastin time (aPTT) at the screening visit
5. Subject with a platelet count below 100×109/L at the screening visit
6. Subject suffering from some acute or chronic medical, surgical or psychiatric significant condition or laboratory abnormality at the screening visit or prior to study treatment administration that, according to Investigator judgement, may increase the risk associated with study participation or study treatment administration, or may interfere with the successful completion or interpretation of the study results
7. Subject with a history of the following: angioedema, cardiac arrhythmia, angina pectoris, myocardial infarction, cerebrovascular accident, cardiac failure, thrombotic events, embolism, coagulopathy, diabetes mellitus, hyperlipidaemia, nephrotic syndrome, acute renal injury, chronic obstructive pulmonary disease, asthma, hepatic disease, reticuloendothelial system dysfunction, or nervous system disorder
8. Subject with known personal or family history of abnormal bleeding episodes
9. Subject not willing to receive study treatment via IM route of administration or unable to receive study treatment via IM route of administration
10. Subject with cardiovascular risk factors based on medical history: active tobacco smoking and/or ongoing diabetes mellitus at the screening visit
11. Subject with thrombosis risk factors: prolonged immobilization within 2 months prior to the screening visit, history of venous or arterial thrombosis, use of estrogens (30 days prior to the study drug administration), indwelling central vascular catheters and hyperviscosity or hypercoagulable states
12. Subject with known history of hypersensitivity/allergic reaction to blood/plasma products
13. Subject with known selective IgA deficiency (with or without antibodies to IgA)
14. Subject who received any plasma-derived product infusion within 12 months prior to study treatment administration
15. Subject who received a blood or plasma transfusion within 12 months prior to study treatment administration
16. Subject with systolic blood pressure >140 mmHg or diastolic blood pressure >90 mmHg at the screening visit and prior to treatment administration
17. Subject with anemia (hemoglobin <12 g/dL in women and 13 g/dL in men) at the screening visit
18. Subjects with proteinuria (>1+ on urine dipstick), blood urea nitrogen (BUN) or creatinine greater than the upper limit of normal at the screening visit
19. Subject with liver enzymes (aspartate aminotransferase [AST], alanine aminotransferase [ALT] and gamma-glutamyl transferase [GGT]) levels greater than the upper limit of normal at screening visit
20. Subject who received any dose of parenteral, oral, or inhaled corticosteroids, immunosuppressants, or immunomodulators within 6 weeks prior to the screening visit
21. Subject who received any live virus vaccine within five months prior to the screening visit
22. Subject not willing to postpone receiving any live virus vaccines until 6 months after receiving IP
23. Currently receiving any anti-viral treatment, regardless of the route of administration
24. Subject with virus safety laboratory results (serology and/or nucleic acid amplification technology [NAT]) indicative of a current infection with hepatitis A virus (HAV), hepatitis B virus (HBV), hepatitis C virus (HCV), human immunodeficiency virus (HIV) or parvovirus B19 (B19V) at the screening visit
25. Participated in another clinical trial within 30 days prior to the screening visit or has received any IPs within 3 months prior to the screening visit
26. Positive urine drug panel testing at the screening visit or prior to study treatment administration
27. Known or suspected abuse of alcohol, opiates, psychotropic agents or other drugs or chemical substances; or has done so in the 12 months prior to the screening visit
28. In the opinion of the Investigator, the subject may have compliance problems with the protocol and the procedures of the protocol
29. Subject who has already been included in a previous group for this clinical study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2017-10-31 (Actual); Primary Completion 2018-04-27 (Actual); Study Completion 2018-07-19 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Vince & Associates Clinical Research, Inc., Overland Park, Kansas, United States

REFERENCES:
- [Derived] Kankam M, Griffin R, Price J, Michaud J, Liang W, Llorens MB, Sanz A, Vince B, Vilardell D. Polyvalent Human Immune Globulin: A Prospective, Open-Label Study Assessing Anti-Hepatitis A Virus (HAV) Antibody Levels, Pharmacokinetics, and Safety in HAV-Seronegative Healthy Subjects. Adv Ther. 2020 May;37(5):2373-2389. doi: 10.1007/s12325-020-01327-9. Epub 2020 Apr 16. PMID 32301062

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 146 subjects were screened for the study, and 8 of them were rescreened. The screen failures were mainly due to body mass index out-of-range. A total of 28 subjects were enrolled in the study.
Period: Overall Study
Arm/Group | Immune Globulin (Human) GamaSTAN
Started | 28
Completed | 26
Not Completed | 2

BASELINE CHARACTERISTICS:
Arm/Group | Immune Globulin (Human) GamaSTAN
Number analyzed (Participants) | 28
Age, Continuous [Mean (Full Range); unit: years] | 41 [22 to 61]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 25
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 9
  White | 18
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects Maintaining Protective Anti- HAV Antibody Levels
Description: Percentage of subjects maintaining anti-HAV antibody levels ≥10 mIU/mL up to Day 60 following study treatment administration.
Time Frame: Day 60
Population: The efficacy analysis was performed using the Evaluable Population.There are 26 subjects in the Evaluable Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Immune Globulin (Human) GamaSTAN
Number analyzed (Participants) | 26
Participants | 26

ADVERSE EVENTS:
Time Frame: Adverse events occurring at any time between signing of the subject's ICF and the last day of the subject's participation in the clinical trial were reported. The total time period for the adverse event data collection was 178 days.
Arm/Group | Immune Globulin (Human) GamaSTAN
All-Cause Mortality (participants affected / at risk) | 0/28
Serious Adverse Events (participants affected / at risk) | 0/28
Other Adverse Events (participants affected / at risk) | 28/28
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Immune Globulin (Human) GamaSTAN (N=28)
Injection site pain (General disorders) | 20 (52)
Vascular access site haemorrhage (Injury, poisoning and procedural complications) | 2 (3)
Neutrophil count decreased (Investigations) | 2 (2)
White blood cell count decreased (Investigations) | 2 (2)
Headache (Nervous system disorders) | 5 (5)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Site may publish results from the Study, after providing Sponsor thirty days' notice prior to submitting a manuscript or other materials related to the Study to any outside party. At Sponsors' request, Site will remove any Confidential Information (other than Study results), and Site will upon Sponsors' request, delay publication or presentation for a period of up to one hundred twenty days to allow Sponsor to protect its interests in any Sponsor Inventions.

DOCUMENTS (2):
  • Study Protocol (2018-01-22): https://cdn.clinicaltrials.gov/large-docs/33/NCT03351933/Prot_000.pdf
  • Statistical Analysis Plan (2018-04-24): https://cdn.clinicaltrials.gov/large-docs/33/NCT03351933/SAP_001.pdf